CLINICAL TRIAL: NCT04414826
Title: Preliminary Efficacy of a One-Session Mindfulness Telehealth Intervention for Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Professor of Psychology, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-04-0088
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Loneliness
Keywords: Loneliness; Mindfulness; Telehealth; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Mindfulness; Methods

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of three groups: (a) Mindfulness alone; (b) Mindfulness + Compassion; and (c) Wait-list control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness + Compassion (MC) Intervention (Active Comparator): Subjects assigned to this condition will participate in an hour-long, one-session telehealth intervention teaching both mindfulness and compassion skills.
  Interventions: Behavioral: Mindfulness + Compassion Intervention (MC)
- Mindfulness Alone (MO) Intervention (Active Comparator): Subjects assigned to this condition will participate in an hour-long, one-session telehealth intervention teaching mindfulness skills alone.
  Interventions: Behavioral: Mindfulness Alone (MO) Intervention
- Waitlist Control (WL) (Placebo Comparator): Those in the wait-list control condition will wait one week and complete a one-week follow-up assessment before being randomized to one of the two intervention conditions.
  Interventions: Behavioral: Mindfulness Alone (MO) Intervention; Behavioral: Mindfulness + Compassion Intervention (MC)

INTERVENTIONS:
Behavioral: Mindfulness Alone (MO) Intervention — Participants will receive a one-session, hour-long telehealth intervention emphasizing awareness and non-reactivity skills.
  Arms: Mindfulness Alone (MO) Intervention; Waitlist Control (WL)
Behavioral: Mindfulness + Compassion Intervention (MC) — Participants will receive a one-session, hour-long telehealth intervention emphasizing awareness, non-reactivity, and compassion skills.
  Arms: Mindfulness + Compassion (MC) Intervention; Waitlist Control (WL)

SUMMARY:
The primary aim of this study is to examine the efficacy of a one-session, hour-long HIPAA-compliant video platform-based mindfulness + compassion telehealth intervention on reducing feelings of loneliness during COVID-19 quarantine. Participants (n=120) currently isolating due to COVID-19 will be randomized to one of three interventions: (a) mindfulness + compassion (MC); (b) mindfulness alone (MO); and (c) waitlist control (WL).

The investigators predict that participants in the active intervention groups (mindfulness or mindfulness + compassion) will show a significantly greater reduction in subjective feelings of loneliness at one week follow-up compared to those in the waitlist control group. Additionally, investigators predict that participants in the active intervention groups will show a significantly greater reduction in stress at one week follow-up compared to those in the waitlist control group. Last, investigators predict that participants in the mindfulness + compassion group will show a significantly greater reduction in subjective feelings of loneliness at the 2-week follow-up follow-up relative to those in the mindfulness only group.

DETAILED DESCRIPTION:
Individuals are currently living in an unprecedented time where they are isolated in their homes for an extended period due to the ongoing coronavirus disease 2019 (COVID-19) pandemic. Feelings of loneliness, or perceived social isolation, have often been cited as accompanying objective social isolation. Prior research has established a link between loneliness and a variety of mental health outcomes including increased depressive symptoms, increased stress reactivity, and increased risk of suicidal thoughts and attempts.

The urgency of the COVID-19 pandemic thus necessitates the investigation of potential short-term interventions for loneliness. Research has suggested that longer-term mindfulness interventions may be effective in mitigating feelings of loneliness and its concomitant mental health outcomes. The proposed study seeks to determine the preliminary efficacy of a one-session mindfulness-based telehealth intervention for loneliness during COVID-19. To increase the potency of this mindfulness-based intervention, the investigators aim to incorporate compassion motivated social engagement.

There is ample evidence that mindfulness alone is an effective intervention method for addressing loneliness. However, inclusion of a compassion component may amplify the effects of an intervention on loneliness because prior research has found that less compassion is associated with greater loneliness. To date, no research has explicitly tested the effect of incorporating compassion into a mindfulness intervention for reducing feelings of loneliness.

ELIGIBILITY:
Inclusion Criteria:

1. Access to the Internet with teleconferencing for the HIPAA-compliant video platform
2. Fluent in English
3. Aged 18 - 70 years old
4. Currently isolating due to COVID-19
5. Endorses loneliness as being among the top three issues impacting their life
6. Demonstrates understanding of the constraints of the intervention (e.g. that it is a single session mindfulness training intervention focused on loneliness).
7. Has access to a private setting for completing the intervention
8. Denies suicidality

Exclusion Criteria:

1. Trauma as a primary concern
2. Significant depression with depression as a primary concern
3. Severe mental illness (e.g. bipolar, schizophrenia, borderline personality disorder)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Revised University of California Los Angeles Loneliness Scale - 8 (ULS-8) | Baseline (Day 0), one-week follow-up (Day 14), two-week follow-up (Day 21)
  Change from baseline in self-reported feelings of loneliness and social isolation. Scores range from 8 to 32, with higher scores indicating higher levels of loneliness.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | Baseline (Day 0), one-week follow-up (Day 14), two-week follow-up (Day 21)
  Change from baseline in self-reported feelings of stress. Scores range from 0 to 40, with higher scores indicating more perceived stress.

OTHER OUTCOMES:
Generalized Anxiety Disorder - 7 (GAD-7) | Baseline (Day 0), one-week follow-up (Day 14), two-week follow-up (Day 21)
  Change from baseline in self-reported anxiety symptoms. Scores range from 0 to 21, with higher scores indicating more severe anxiety.
Personal Health Questionnaire Depression Scale - 8 (PHQ-8) | Baseline (Day 0), one-week follow-up (Day 14), two-week follow-up (Day 21)
  Change from baseline in self-reported depressive symptoms. Scores range from 0 to 24, with higher scores indicating higher depressive symptom severity.
Brunnsviken Brief Quality of Life Scale (BBQ) | Baseline (Day 0), one-week follow-up (Day 14), two-week follow-up (Day 21)
  Change from baseline in self-reported quality of life. Scores range from 0 to 48, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Telch, PhD, Study Director — The University of Texas at Austin; Mikael Rubin, MA, Principal Investigator — The University of Texas at Austin
Locations (1):
- Laboratory for the Study of Anxiety Disorders, University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, Analytic Code
Access Criteria: Data will be made available on osf
URL: https://osf.io/hxj2z/

REFERENCES:
- [Background] Shankar A, McMunn A, Banks J, Steptoe A. Loneliness, social isolation, and behavioral and biological health indicators in older adults. Health Psychol. 2011 Jul;30(4):377-85. doi: 10.1037/a0022826. PMID 21534675
- [Background] Cacioppo JT, Hughes ME, Waite LJ, Hawkley LC, Thisted RA. Loneliness as a specific risk factor for depressive symptoms: cross-sectional and longitudinal analyses. Psychol Aging. 2006 Mar;21(1):140-51. doi: 10.1037/0882-7974.21.1.140. PMID 16594799
- [Background] VanderWeele TJ, Hawkley LC, Thisted RA, Cacioppo JT. A marginal structural model analysis for loneliness: implications for intervention trials and clinical practice. J Consult Clin Psychol. 2011 Apr;79(2):225-35. doi: 10.1037/a0022610. PMID 21443322
- [Background] Heinrich LM, Gullone E. The clinical significance of loneliness: a literature review. Clin Psychol Rev. 2006 Oct;26(6):695-718. doi: 10.1016/j.cpr.2006.04.002. Epub 2006 Jun 19. PMID 16952717
- [Background] Creswell JD, Irwin MR, Burklund LJ, Lieberman MD, Arevalo JM, Ma J, Breen EC, Cole SW. Mindfulness-Based Stress Reduction training reduces loneliness and pro-inflammatory gene expression in older adults: a small randomized controlled trial. Brain Behav Immun. 2012 Oct;26(7):1095-101. doi: 10.1016/j.bbi.2012.07.006. Epub 2012 Jul 20. PMID 22820409
- See also: Website for the Laboratory for the Study of Anxiety Disorders — http://UTanxiety.com